CLINICAL TRIAL: NCT05540301
Title: Effectiveness of Modified Sleeper Stretch And Modified Cross-Body Adduction Stretch To Increase Shoulder Internal Rotation Range of Motion In Tennis Players
Brief Title: Sleeper's and Adduction Stretch to Increase Shoulder ROM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King Saud University (Other)
Responsible Party: Principal Investigator, Masood Khan, Principal Investigator, King Saud University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 3/2015/MPT
Record Dates: First submitted 2022-09-11; First posted 2022-09-14 (Actual); Last update posted 2022-09-14 (Actual); Status verified 2022-09

CONDITIONS: Stiffness of Shoulder, Not Elsewhere Classified
Keywords: Sleeper Stretch; Cross-Body Stretch; Range of Motion; Shoulder; Tennis Players

STUDY DESIGN:
Intervention Model Description: Two-group two-factor research design was used.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Modified Sleeper Stretch Group (Experimental): Modified sleeper stretch was performed for four weeks.
  Interventions: Other: Modified sleeper stretching
- Modified Cross-Body Adduction Stretch Group (Active Comparator): Modified cross-body adduction stretch was performed for four weeks.
  Interventions: Other: Modified cross-body adduction stretch

INTERVENTIONS:
Other: Modified sleeper stretching — Modified sleeper stretching was performed on shoulder joint to increase internal rotation range of motion.
  Arms: Modified Sleeper Stretch Group
Other: Modified cross-body adduction stretch — Modified cross-body adduction stretching was performed on shoulder joint to increase internal rotation range of motion.
  Arms: Modified Cross-Body Adduction Stretch Group

SUMMARY:
The study aimed to compare the efficacy of modified sleeper stretch and modified cross-body adduction stretch in improving shoulder internal rotation range of motion and upper limb function. Thirty male lawn tennis players aged between 20 to 35, with more than 150 glenohumeral internal rotation deficiency (GIRD) on the dominant shoulder (compared to the nondominant side) participate in the study and divided into two groups (A and B). Group A received a modified sleeper stretch and group B received a modified cross-body adduction stretch for four weeks, five times per week. The outcome measures were the internal rotation range of motion measured by a universal goniometer and upper limb functions measured by the Disability of the Arm, Shoulder, and Hand (DASH) scale.

ELIGIBILITY:
Inclusion Criteria:

* Lawn Tennis Players
* Male
* more than 15 degree glenohumeral internal rotation deficiency

Exclusion Criteria:

* systemic or metabolic disorders
* a positive test for labral lesions or rotator cuff tears
* a history of recent fracture
* a history of orthopaedic surgery in the upper limbs or cervical region

Ages: 20 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2016-03-08 (Actual); Primary Completion 2017-01-23 (Actual); Study Completion 2017-04-06 (Actual)

PRIMARY OUTCOMES:
Internal rotation range of motion | 4 weeks.
  Internal rotation range of motion (ROM) was measured using the universal goniometer before and after the completion of the intervention. The greater the ROM, the better the prognosis.
Upper limb functions | 4 weeks.
  The Disability of the Arm, Shoulder, and Hand (DASH) scale was used to assess the upper limb functions. The DASH consists mainly of a 30-item disability/symptom scale, scored 0 (no disability) to 100. The higher the score, the worse the prognosis.

CONTACTS AND LOCATIONS:
Overall Officials: Masood Khan, M.P.Th, Principal Investigator — King Saud University
Locations (1):
- King Saud University, Riyadh, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No